CLINICAL TRIAL: NCT04039685
Title: The Effects of Chronic Exercise on UCP1 Gene in Human White Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 4. Browning of WAT
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Obese; Obesity
Keywords: uncoupling protein 1; uncoupling protein one; resistance exercise; aerobic exercise; browning formation; white fat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic exercise group (Experimental)
  Interventions: Other: Effects of an eight weeks aerobic exercise followed by an eight weeks de-training period on UCP1 gene of human white adipose tissue
- Resistance exercise group (Experimental)
  Interventions: Other: Effects of an eight weeks resistance exercise followed by an eight weeks de-training period on UCP1 gene of human white adipose tissue
- Combined (aerobic+resistance) exercise group (Experimental)
  Interventions: Other: Effects of an eight weeks combined (aerobic+resistance) exercise followed by an eight weeks de-training period on UCP1 gene of human white adipose tissue
- Non-exercise group (No Intervention)

INTERVENTIONS:
Other: Effects of an eight weeks aerobic exercise followed by an eight weeks de-training period on UCP1 gene of human white adipose tissue — The investigators evaluated the effects of an eight weeks aerobic exercise program and a following of eight weeks of a de-training period on UCP1 gene in previously non-regular exercisers healthy adult men
  Arms: Aerobic exercise group
Other: Effects of an eight weeks resistance exercise followed by an eight weeks de-training period on UCP1 gene of human white adipose tissue — The investigators evaluated the effects of an eight weeks resistance exercise program and a following of eight weeks of a de-training period on UCP1 gene in previously non-regular exercisers healthy adult men
  Arms: Resistance exercise group
Other: Effects of an eight weeks combined (aerobic+resistance) exercise followed by an eight weeks de-training period on UCP1 gene of human white adipose tissue — The investigators evaluated the effects of an eight weeks combined (aerobic+resistance) exercise program and a following of eight weeks of a de-training period on UCP1 gene in previously non-regular exercisers healthy adult men
  Arms: Combined (aerobic+resistance) exercise group

SUMMARY:
Obesity is characterized by excessive white adipose tissue (WAT) that increases risk for disease. About 700 million adults are obese worldwide, designating the need of reducing excessive WAT in humans and subsequently the risk for disease. For this reason, previous research focused on the thermogenic capacity of white adipocytes in response to chronic exercise. It is suggested that the latter occurs due to increased demand of oxidation during exercise to maintain non-esterified fatty acids flux in the circulation, thus to maintain energy supply White adipocytes express the uncoupling protein one (UCP1), which dissipates chemical energy in the mitochondria to produce heat in response to cold exposure. UCP1 was thought that exclusively appears in brown adipose tissue (BAT), which during the mitochondrial electron transport chain process, bypasses the adenosine triphosphate (ATP) synthase to produce heat, as a thermoregulatory mechanism of maintaining body temperature. Its presence in white adipocytes, indicates a thermogenic capacity of WAT, which could lead to similar health benefits as those reported for increased BAT activity; mainly reduced body mass index (BMI) and fat mass, which designate body weight loss and reduced obesity phenotype.

The investigators aimed to identify whether UCP1 in human WAT is altered by chronic exercise.

DETAILED DESCRIPTION:
The investigators obtained three (baseline, post-exercise, post-de-training) subcutaneous fat biopsies from 32 healthy men who undertook three different eight week exercise programs [aerobic (9 participants), resistance (8 participants), combined (aerobic+resistance, 8 participants)] and a non-exercise group (7 participants), followed by an eight week de-training period. Exercise intensity was set at 65% of peak oxygen consumption (VO2peak) and 1 repetition maximum (1RM) throughout the exercise period, while the content of the exercise programs based on a previous study that examined the PGC1a gene, which is thought that increases UCP1 in human white adipose tissue (WAT). Exercise performed in three local gyms in Trikala, Thessaly, Greece, each for every exercise group to avoid cross-contamination between participants, while the exercise supervisors were blinded to the aim of the study. Measurements for anthropometry, body composition, resting energy expenditure (REE), and subcutaneous fat biopsy were obtained at baseline, post-exercise (week 8) and post de-training (week 16) periods while diet data were randomly collected for two weekdays and one weekend day at baseline, 8th and 16th week. VO2peak and 1RM were measured at baseline, 4th (to adjust the required exercise intensity at 65%), 8th and 16th week.

Anthropometry The participants visited the laboratory between 07:00 and 09:00 am and the following anthropometry measures took part: Height was measured using a Seca (Hamburg, Germany) device and weight using a scale (KERN & Sohn GmbH, Version 5.3, Germany) while waist-to-hip ratio was measured using a tape measure and blood pressure through an acoustic method using an Aneroid sphygmomanometer. Percent body fat and fat-free mass were measured via bioelectrical impedance using a body composition monitor (Fresenius Medical Care AG & Co. KGaA D-61346 Bad Hamburg, Germany).

Fat biopsies All biopsies were executed by an experienced surgeon following a previous methodology via a non-diathermy method. The participants underwent a subcutaneous fat biopsy after at least an eight hour fast and they were instructed to refrain from exercise, alcohol, and passive smoking in 72 hours prior the biopsy procedure in order to minimize the risk for misleading results. Each participant was positioned on a surgical bed in a supine position. The site of the incision was disinfected and a 10 ml of xylocaine 2%-no adrenaline was injected in the region of the incision for local anaesthesia. An incision on the skin and subcutaneous tissue until adipose tissue was revealed, was executed approximately 3-5 centimetres nearby the navel while the incision length was approximately 2-2.5 centimetres. Subsequently, the subcutaneous tissue was removed with an operating scissors and when the adipose tissue became visible nearly 500 milligrams of adipose tissue was captured and removed. The collected adipose tissue was immediately immersed in liquid nitrogen of -190° Celsius. For the final deposition the samples were placed in Eppendorfs and they were deposited in a freezer at -80° Celsius until analyses.

UCP1 mRNA analysis The investigators who performed the gene and protein expression analyses were blinded to the aim of the study. Total RNA was extracted from adipose tissue biopsies using RNeasy Lipid Tissue mini kit (QIAGEN) following the manufacturer's protocol. First-strand cDNAs were synthesized from equal amounts of total RNA using random primers and M-MLV reverse transcriptase (Promega). Quantitative real time polymerase chain reaction for the UCP1 gene was performed using Sybr Green fluorophore. The change in fluorescence at every cycle was monitored and a threshold cycle above background for each reaction was calculated. A melt curve analysis was performed following every run to ensure a single amplified product for every reaction. All reactions were carried out in at least duplicated for every sample. 18S rRNA gene was constantly expressed under all experimental conditions and was then used as a reference gene for normalization given that this gene was suggested as the most appropriate one for normalization of UCP1 mRNA.

UCP1 protein analysis Subcutaneous adipose tissue was homogenized in RIPA Lysis Buffer with protease inhibitors (Sigma-Aldrich, Milan, Italy), centrifuged at 800g for 10 minutes at 4° Celsius and then the middle layer was collected. Equal amounts (50 micrograms) of proteins were separated on 10% SDS-polyacrylamide gel, transferred to a nitrocellulose membrane. UCP1 from subcutaneous adipose tissue samples were detected by primary antibodies, respectively rabbit polyclonal anti-human UCP1 (1:1000, Sigma-Aldrich, Milan, Italy) and mouse monoclonal anti-human β-actin (1:5000, Sigma-Aldrich, Milan, Italy). Secondary antibodies were peroxidase-conjugated anti-rabbit IgG for UCP1 and anti-mouse IgG for β-actin. Human adipocytes that treated with 100uM menthol were used as positive controls for UCP1 protein expression according to previous methodology. Western blotting analysis was performed using Immobilion Western Chemiluminescent HRP Substrate (Millipore) and detection was made using photographic films. The images have been analysed by densitometry, which evaluates the relative amount of protein staining and quantifies the results in terms of optical density.

REE assessments REE assessments were conducted between 07:00 to 09:00 am following 12 hours of fast, while participants refrained from exercise, alcohol, and passive smoking in 72 hours prior to the measurements. REE was measured using an automated gas analyzer (Vmax, CareFusion, USA) that was attached to the participants to record respiratory variables every 20 seconds in a supine position for 30 minutes in a quiet room of 22-24° Celsius. From the 30 minutes of the collected data, the first and last five minutes were removed. Finally, the remaining 20 minutes of the collected data were averaged to obtain the final REE (calories) value. Respiratory gas measurements were extracted using the Weir equation to convert VO2 and VCO2 values to REE (calories) values. To ensure accuracy of the REE measurements the average respiratory exchange ratio was also verified according to previous methodology.

VO2peak and 1RM assessments At baseline, a pre-screening was performed for each participant to identify their eligibility to undertake a VO2peak test using the Physical Activity Readiness Questionnaire. To ensure the familiarization of the participants with the VO2peak test a detailed verbal description of the protocol was given in advance. The protocol involved a five minute warm-up and a familiarization period of a cycling in a Monark Ergomedic 839E, Vansbro, Sweden. Consequently, the test involved a three minute of pedaling at 60 revolutions per minute at 60 Watts followed by an increment of 30 Watts/minute until volitional exhaustion. An automated gas analyzer (Vmax, CareFusion, USA) was attached to the participants to record respiratory variables every 20 seconds. The highest oxygen uptake (milliliters/minute) for any 20 second interval was recorded as the final VO2peak value.

The 1RM of leg extension and chest press were tested as following: A suitable weight was adjusted for each participant in order to not be able to lift it for no more than 10 repetitions. The number of the repetitions were then calculated and a norm was used to predict the 1RM using the weight in kilograms that each participant lifted and the number of the repetitions that were performed.

Diet assessment Participants were randomly contacted by telephone - by an independent assistant who was blinded to the aim of the study - on three separate days (two weekdays, one weekend day) during a week period for the completion of a three-day diet record. All food and beverages consumed on the day of contact were recorded. Three-day diet records were collected at baseline, 8th and 16th week of the intervention. All diet records were analyzed by another trained assistant who was blinded to the aim of the study using Nutritionist Pro, Version 5.4.0, Axxya Systems (Redmond, WA, USA). This software (i.e. Nutritionist Pro) has been previously used for research purposes. For the analysis, a search was conducted in Nutritionist Pro for each food and beverage consumed. Details regarding the amount and preparation of each food and/or beverage were also included. Once all the relevant information regarding the food or beverage was entered into the software, a corresponding list of macro and micro-nutrient content was provided and subsequently saved. This process was repeated for all food and beverages listed on the diet record. If a particular food or beverage was not found within the Nutritionist Pro database, the investigator manually entered the macro and micro-nutrient content of that particular food and saved it to the database for future use. The feedback provided by the software for each food or beverage included the following dietary variables: total energy intake (calories), weight of food (grammars), protein (grammars), carbohydrate (grammars), total fat (grammars), total sugar (grammars) and caffeine (micro-grammars).

ELIGIBILITY:
Inclusion Criteria:

* adult men
* healthy
* no chronic disease
* no medication treatment
* no regular exercisers

Exclusion Criteria:

* women
* non-adult men
* chronic disease individuals
* any medication treatment
* acute illness
* regular exercisers

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
UCP1 mRNA expression in white adipocytes | Baseline measurements; measurements at the end of the exercise intervention (8th week); measurements at the end of the de-training period (16th week)
  UCP1 mRNA expression was measured via fat biopsy samples from the subcutaneous abdominal area at baseline, at the end of the exercise intervention (8th week) and at the end of the de-training period (16th week)
UCP1 protein concentration in white adipocytes | Baseline measurements; measurements at the end of the exercise intervention (8th week); measurements at the end of the de-training period (16th week)
  UCP1 protein concentration was measured via fat biopsy samples from the subcutaneous abdominal area at baseline, at the end of the exercise intervention (8th week) and at the end of the de-training period (16th week)

CONTACTS AND LOCATIONS:
Locations (1):
- Petros Dinas, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided